CLINICAL TRIAL: NCT00200057
Title: Medtronic InterStim® Sacral Nerve Stimulation Therapy for Bowel Control: Fecal Incontinence Study
Brief Title: Sacral Nerve Stimulation Therapy for the Treatment of Chronic Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sudha Iyer, Clinical Research Manager, Medtronic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G010206
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2011-08-30 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence; InterStim
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: InterStim Sacral Nerve Stimulation Therapy — Open label study. All subjects that qualify for the study will be implanted.

SUMMARY:
Fecal incontinence (FI) is a difficulty in storing gas, liquid stool or solid stool (bowel movement) in order to expel it at a proper time and place. Patients who suffer from FI may experience passive FI (difficulty in sensing stool in the rectum) or urgency (able to sense a bowel movement but cannot hold the stool until an acceptable time and place). FI is not a life-threatening disease, but it is often profoundly distressing and socially incapacitating.

If a patient is suffering with symptoms of chronic FI despite trying oral medications, biofeedback and/or other more conservative treatments, a patient may be eligible to participate in a clinical research study to evaluate the safety and effectiveness of sacral nerve stimulation for the treatment of chronic fecal incontinence. One hundred-twenty (120) patients will be implanted with medical devices and followed closely for twelve months, and then once a year after that until the study closes. There are up to 20 centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* 18 years of age or older.
* Patient is diagnosed with chronic fecal incontinence of a duration greater than 6 months (>12 months post-vaginal childbirth) and defined as > 2 incontinent episodes on average per week of more than staining recorded during the baseline diary period.
* Failed or are not candidates for more conservative treatments.
* Willing and competent to completely and accurately fill out bowel diaries and questionnaires throughout the study.

Exclusion Criteria:

* Congenital anorectal malformations.
* Active participation in another bowel disorder investigational study.
* Present rectal prolapse.
* Previous rectal surgery (such as rectopexy or resection) or sphincteroplasty done < 12 months prior to study enrollment (24 months for cancer).
* Neurological diseases such as clinically significant peripheral neuropathy or complete spinal cord injury (i.e. paraplegia).
* Grade III hemorrhoids.
* Known or suspected organic disorders of the bowel (i.e. Inflammatory bowel disease such as Crohn's or ulcerative colitis).
* Chronic watery diarrhea, unmanageable by drugs or diet, as primary cause of fecal incontinence. (Incontinent episodes with a Bristol stool consistency of > 6 for > 4 days during the baseline diary period will be exclusionary, unless the investigator determines that the diary is not indicative of chronic watery diarrhea.)
* Pregnancy or planned pregnancy.
* Patients for whom patient materials are not available in a language understood by the patient.
* Life expectancy of less than one year.
* Patient characteristics indicating a poor understanding of the study or poor compliance with the study protocol (i.e., patients unable to adequately operate equipment, patients unwilling or unable to return for scheduled follow-up visits).
* Patients with a history of pelvic irradiation who present with visible or functional effects of irradiation.
* Patients with active anal abscesses or fistulas.
* Patients with anatomical limitations that would prevent the successful placement of an electrode.
* Patients with knowledge of planned MRIs, diathermy, microwave, or RF energy.
* Patients with other implantable neurostimulators, pacemakers or defibrillators.
* Defect of external anal sphincter of >60 degrees or amenable to surgical repair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2002-01; Primary Completion 2007-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudha Iyer, PhD, Study Director — Medtronic
Locations (13):
- United States (12):
  - Contact Medtronic for specific site information, Los Angeles, California
  - Contact Medtronic for specific site information, San Francisco, California
  - Contact Medtronic for specific site information, Washington D.C., District of Columbia
  - Contact Medtronic for specific site information, Weston, Florida
  - Contact Medtronic for specific site information, Chicago, Illinois
  - Contact Medtronic for specific site information, Kansas City, Kansas
  - Contact Medtronic for specific site information, New Orleans, Louisiana
  - Contact Medtronic for specific site information, Burlington, Massachusetts
  - Contact Medtronic for specific site information, Minneapolis, Minnesota
  - Contact Medtronic for specific site information, Cleveland, Ohio
  - Contact Medtronic for specific site information, Oklahoma City, Oklahoma
  - Contact Medtronic for specific site information, Fort Worth, Texas
- Contact Medtronic for specific site information, Fleurimont, Quebec, Canada

REFERENCES:
- [Result] Wexner SD, Coller JA, Devroede G, Hull T, McCallum R, Chan M, Ayscue JM, Shobeiri AS, Margolin D, England M, Kaufman H, Snape WJ, Mutlu E, Chua H, Pettit P, Nagle D, Madoff RD, Lerew DR, Mellgren A. Sacral nerve stimulation for fecal incontinence: results of a 120-patient prospective multicenter study. Ann Surg. 2010 Mar;251(3):441-9. doi: 10.1097/SLA.0b013e3181cf8ed0. PMID 20160636
- [Result] Wexner SD, Hull T, Edden Y, Coller JA, Devroede G, McCallum R, Chan M, Ayscue JM, Shobeiri AS, Margolin D, England M, Kaufman H, Snape WJ, Mutlu E, Chua H, Pettit P, Nagle D, Madoff RD, Lerew DR, Mellgren A. Infection rates in a large investigational trial of sacral nerve stimulation for fecal incontinence. J Gastrointest Surg. 2010 Jul;14(7):1081-9. doi: 10.1007/s11605-010-1177-z. Epub 2010 Mar 31. PMID 20354809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical investigation began on January 14, 2002, and the first implant occurred on May 03, 2002. The study was closed to enrollments on June 15, 2006, and the last implant occurred on August 04, 2006.
Pre-assignment Details: All patients who signed an informed consent were considered enrolled in the study. Of the 285 subjects who enrolled in the study, 132 subjects underwent acute test stimulation with 129 proceeding to the sub-chronic test stimulation phase. Of these, 120 subjects qualified for permanent implant. All 120 patients were successfully implanted.
Groups:
- Implanted Subjects: Subjects implanted with Sacral Nerve Stimulation (SNS) device.
Period: Overall Study
Arm/Group | Implanted Subjects
Started | 120
1 Month Follow-up | 117
3 Month Follow-up | 116
6 Month Follow-up | 114
12 Month Follow-up | 111
Completed | 111
Not Completed | 9
Not completed — Lack of Efficacy | 3
Not completed — Exited due to terminal illness of PI | 2
Not completed — Withdrawal by Subject | 1
Not completed — Change in medical condition | 1
Not completed — Infection | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 60.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 87
  Canada | 19
  Australia | 14
Weekly Fecal Incontinent Episodes [Mean (Standard Deviation); unit: incontinent episodes per week] — A bowel diary was used by subjects to record information about their bowel elimination frequency. Over the 14-day diary period, subjects recorded the date and time of each bowel episode and responded to questions related to each bowel episode, including amount of incontinence (none, staining, minor soiling, major soiling) and urgency (no, yes). A bowel movement was considered incontinent if the amount of incontinence was minor or major soiling.
  incontinent episodes per week | 9.39 (7.27)
Weekly Fecal Incontinent Days [Mean (Standard Deviation); unit: incontinent days per week] — A bowel diary was used by subjects to record information about their bowel elimination frequency. Over the 14-day diary period, subjects recorded the date and time of each bowel episode and responded to questions related to each bowel episode, including amount of incontinence (none, staining, minor soiling, major soiling) and urgency (no, yes). A bowel movement was considered incontinent if the amount of incontinence was minor or major soiling. A day in a diary period was considered as an incontinent day if there was at least one incontinent episode during that day.
  incontinent days per week | 4.51 (1.61)
Weekly Urgent Fecal Incontinent Episodes [Mean (Standard Deviation); unit: urgent incontinent episodes per week] — A bowel diary was used by subjects to record information about their bowel elimination frequency. Over the 14-day diary period, subjects recorded the date and time of each bowel episode and responded to questions related to each episode, including amount of incontinence (none, staining, minor soiling, major soiling) and urgency (no, yes). A bowel movement was considered incontinent if the amount of incontinence was minor or major soiling. A bowel movement was considered urgent if the answer to the urgency question was yes and it was associated with incontinence.
  urgent incontinent episodes per week | 4.95 (4.88)
Fecal Incontinence Quality of Life (FIQOL) Scale 1 - Lifestyle [Mean (Standard Deviation); unit: units on a scale] — Baseline measure from all subjects who were successfully implanted and completed the Fecal Incontinence Quality of Life (FIQOL) at baseline, n=119. Scales range from 1 to 5, with a 1 indicating a lower functional status of quality of life.
  units on a scale | 2.31 (0.85)
FIQOL Scale 2 - Coping/Behavior [Mean (Standard Deviation); unit: units on a scale] — Baseline measure from all subjects who were successfully implanted and completed the FIQOL at baseline, n=119. Scales range from 1 to 5, with a 1 indicating a lower functional status of quality of life.
  units on a scale | 1.49 (0.53)
FIQOL Scale 3 - Depression/Self-Perception [Mean (Standard Deviation); unit: units on a scale] — Baseline measure from all subjects who were successfully implanted and completed the FIQOL at baseline, n=119. Scales range from 1 to 5, with a 1 indicating a lower functional status of quality of life.
  units on a scale | 2.53 (0.81)
FIQOL Scale 4 - Embarrassment [Mean (Standard Deviation); unit: units on a scale] — Baseline measure from all subjects who were successfully implanted and completed the FIQOL at baseline, n=119. Scales range from 1 to 5, with a 1 indicating a lower functional status of quality of life.
  units on a scale | 1.60 (0.63)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With at Least 50% Reduction in Number of Incontinent Episodes Per Week
Description: The primary efficacy objective was to demonstrate that at least 50% of subjects will achieve at least 50% reduction in the number of fecal incontinent episodes per week at 12 months post-implant compared to baseline. Subjects who achieve at least 50% reduction in the number of fecal incontinent episodes per week at 12 months post-implant compared to baseline are considered "successes."
  The observed therapeutic success rate is calculated as the proportion of implanted subjects who achieve at least 50% reduction in the number of incontinent episodes per week from baseline to twelve months.
Time Frame: Baseline and 12 months
Population: All subjects who were successfully implanted were included in the analysis. A modified worst-case analysis was used for missing data, where all subjects who were missing 12-month data were classified as failures, unless there was a subsequent diary available, in which case the subsequent diary was substituted for the missing 12-month data.
Measure: Mean (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 120
proportion of subjects | 0.73 [0.64 to 0.81]
Statistical Analysis 1: Comparison: Implanted Subjects; The exact Binomial test (two-sided) for one-sample proportions was used to test the null hypothesis that the success rate is equal to 0.5; Test type: Superiority or Other; p < 0.0001, Exact Binomial — No multiplicity adjustments were made for the primary outcome analysis. Two-tailed p-values were considered statistically significant if they were less than 0.05; Proportion = 0.73, 95% CI 2-sided [0.64 to 0.81]

2. Secondary Outcome: Proportion of Subjects With at Least 50% Reduction in Number of Incontinent Days Per Week
Description: This secondary objective was to demonstrate that at least 50% of subjects achieved at least 50% reduction in the number of incontinent days per week at 12 months post-implant compared to baseline. Subjects who achieve at least 50% reduction in the number of fecal incontinent days per week at 12 months post-implant compared to baseline are considered "successes."
  The observed therapeutic success rate is calculated as the proportion of implanted subjects who achieve at least 50% reduction in the number of incontinent days per week from baseline to twelve months.
Time Frame: Baseline and 12 months
Population: All subjects who were successfully implanted were included in the analysis. A modified worst-case analysis was used for missing data, where all subjects who were missing 12-month data were classified as failures unless there was a subsequent diary available, in which case the subsequent diary was substituted for the missing 12-month data.
Measure: Mean (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 120
proportion of subjects | 0.73 [0.64 to 0.81]
Statistical Analysis 1: Comparison: Implanted Subjects; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Exact Binomial — The Hochberg procedure for multiplicity adjustment was used for all secondary objectives; Proportion = 0.73, 95% CI 2-sided [0.64 to 0.81]

3. Secondary Outcome: Change in Quality of Life From Baseline to 12 Months: Scale 1 - Lifestyle
Description: This secondary efficacy objective was to demonstrate improvement in Fecal Incontinence Quality of Life (FIQOL) scores at 12 months post-implant compared to baseline. Scales range from 1 to 5, with a 1 indicating a lower functional status of quality of life. The four component scales of the FIQOL instrument were evaluated separately.
Time Frame: Baseline and 12 months
Population: All subjects who were successfully implanted were included in the analysis. The modified worst-case analysis was used to account for subjects who did not complete the FIQOL questionnaire at either baseline or 12 months; these subjects were classified as no change from baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 120
units on a scale | 0.92 (0.92)
Statistical Analysis 1: Comparison: Implanted Subjects; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The Hochberg procedure for multiplicity adjustment was used for all secondary objectives

4. Secondary Outcome: Change in Quality of Life From Baseline to 12 Months: Scale 2 - Coping/Behavior
Description: as for outcome 3
Time Frame: Baseline and 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 120
units on a scale | 1.12 (0.99)
Statistical Analysis 1: Comparison: Implanted Subjects; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The Hochberg procedure for multiplicity adjustment was used for all secondary objectives

5. Secondary Outcome: Change in Quality of Life From Baseline to 12 Months: Scale 3 - Depression/Self-Perception
Description: as for outcome 3
Time Frame: Baseline and 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 120
units on a scale | 0.86 (0.96)
Statistical Analysis 1: Comparison: Implanted Subjects; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The Hochberg procedure for multiplicity adjustment was used for all secondary objectives

6. Secondary Outcome: Change in Quality of Life From Baseline to 12 Months: Scale 4 - Embarrassment
Description: as for outcome 3
Time Frame: Baseline and 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 120
units on a scale | 1.06 (1.00)
Statistical Analysis 1: Comparison: Implanted Subjects; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The Hochberg procedure for multiplicity adjustment was used for all secondary objectives

7. Secondary Outcome: Proportion of Subjects With at Least 50% Reduction in Number of Urgent Incontinent Episodes Per Week
Description: This secondary objective was to demonstrate that at least 50% of subjects achieved at least 50% reduction in the number of urgent incontinent episodes per week at 12 months post-implant compared to baseline. Subjects who achieve at least 50% reduction in the number of urgent fecal incontinent episodes per week at 12 months post-implant compared to baseline are considered "successes."
  The observed therapeutic success rate is calculated as the proportion of implanted subjects who achieve at least 50% reduction in the number of urgent incontinent episodes per week from baseline to 12 months.
Time Frame: Baseline and 12 months
Population: All subjects who were successfully implanted were included in this analysis. The modified worst-case analysis for missing data was used, so that all subjects with missing 12-month data were classified as failures, unless there was a subsequent diary available, in which case the subsequent diary was substituted for the missing 12-month data.
Measure: Mean (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 120
proportion of subjects | 0.71 [0.62 to 0.79]
Statistical Analysis 1: Comparison: Implanted Subjects; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Exact Binomial — The Hochberg procedure for multiplicity adjustment was used for all secondary objectives; Proportion = 0.71, 95% CI 2-sided [0.62 to 0.79]

ADVERSE EVENTS:
Time Frame: One hundred twenty subjects were implanted with the InterStim system, accumulating 2758 device months of experience (ranging from 2.2 to 61 months, averaging 23 months) through the data cutoff date of May 27, 2008.
Description: Adverse events listed below were collected after permanent implant of the device through the data cutoff date.
Arm/Group | Implanted Subjects
Serious Adverse Events (participants affected / at risk) | 41/120
Other Adverse Events (participants affected / at risk) | 88/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted Subjects (N=120)
Implant site infection (Infections and infestations) | 5 (5)
Urinary tract infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Perianal abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Eating disorder (Psychiatric disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (3)
Carotid artery occlusion (Nervous system disorders) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Varicose vein (Vascular disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 5 (7)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (3)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Volvulus of bowel (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Implant site pain (General disorders) | 4 (4)
Therapeutic product ineffective (General disorders) | 1 (1)
Implant site erosion (General disorders) | 1 (1)
Ulcer (General disorders) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Lead migration/dislodgment (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted Subjects (N=120)
Implant site infection (Infections and infestations) | 8 (8)
Urinary tract infection (Infections and infestations) | 8 (10)
Insomnia (Psychiatric disorders) | 6 (6)
Paraesthesia (Nervous system disorders) | 13 (16)
Faecal incontinence (Gastrointestinal disorders) | 29 (35)
Diarrhoea (Gastrointestinal disorders) | 16 (20)
Proctalgia (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 7 (7)
Haemorrhoids (Gastrointestinal disorders) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (11)
Urinary incontinence (Renal and urinary disorders) | 14 (14)
Implant site pain (General disorders) | 28 (33)
Pain (General disorders) | 8 (8)
Laboratory test abnormal (Investigations) | 8 (13)
Change in sensation of stimulation (General disorders) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No